CLINICAL TRIAL: NCT00237497
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Ramelteon Compared to Placebo With Zopiclone as a Reference Arm in Adults With Chronic Insomnia
Brief Title: Safety and Efficacy of Ramelteon in Adults With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375-EC301; U1111-1114-1542 (Registry Identifier: WHO); 2004-004350-91 (EudraCT Number)
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Balance
Keywords: Insomnia; Center of Pressure; Postural Sway; Drug Therapy; Balance and Stability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon; zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Zopiclone 7.5 mg QD (Active Comparator)
  Interventions: Drug: Zopiclone
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily for up to 28 nights.
  Other Names: Rozerem; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Zopiclone — Zopiclone 7.5 mg, tablets, orally, once daily for up to 28 nights.
  Other Names: Zimovane; Imovane; Rovane
  Arms: Zopiclone 7.5 mg QD
Drug: Placebo — Placebo-matching tablets, orally, once daily for up to 28 nights.
  Arms: Placebo QD

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Ramelteon, once daily (QD), compared to placebo with Zopiclone in adults with chronic insomnia

DETAILED DESCRIPTION:
A vast majority of people are affected by chronic insomnia in the western world. Several studies have looked at this and have estimated that 30% to 48% of the general population is affected at some time in their life with a form of insomnia that goes on for several months, and about one third of those are described as severely affected. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia-related conditions that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism, and greater rates of accidents.

This study will examine the effect of ramelteon on balance/postural stability on Night 14 at peak plasma concentration levels, compared with placebo and using zopiclone as the reference arm.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 64 years, inclusive.
* Capable of understanding and willing to comply with the protocol and had to fully understand and sign the informed consent document at screening prior to any study-related procedures being performed.

In addition, subjects had to meet the following study-specific criteria:

* Chronic insomnia as defined by:

  * A complaint of difficulty initiating or maintaining sleep or of nonrestorative sleep that lasted for at least 3 months.
  * The sleep disturbance (or associated daytime fatigue) caused clinically significant distress or impairment in social, occupational, or other important areas of functioning.
  * The disturbance did not occur exclusively during the course of narcolepsy, breathing related sleep disorder, circadian rhythm sleep disorder or a parasomnia.
  * The sleep disturbance did not occur exclusively during the course of another mental disorder (eg, major depressive disorder, generalized anxiety disorder, a delirium).
  * The disturbance was not due to the direct physiological effects of a substance (eg, a drug of abuse, a medication) or a general medical condition.
* Based on sleep history, a subjective sleep latency (sSL) ≥45 minutes.
* Based on sleep history, a subjective total sleep time (sTST) ≤6.5 hours.
* Based on sleep history, a mean LPS of ≥20 minutes on 2 consecutive screening nights with neither night <15 minutes.
* Based on sleep history, their habitual bedtime was between 10:00 PM and 1:00 AM.
* Able to stand with eyes closed, arms at side and feet apart at hips width for at least 1 minute with out taking a step.
* A body mass index (BMI) between 18 and 34, inclusive.
* Used pharmacological assistance to sleep 0 to 4 times per week in the last 3 months.
* Agreed to discontinue use of all pharmacological sleep aids 1 week prior to the dose of singleblind study medication and throughout the entire duration of the study.
* Women of childbearing potential were non-pregnant and non-lactating and had appropriate birth control (barrier methods, hormonal contraceptives, and/or intrauterine devices) for the entire duration of the study (women who were not of childbearing potential were postmenopausal for 1 year or had a history of hysterectomy and/or bilateral oophorectomy).

Exclusion Criteria:

* A known hypersensitivity to ramelteon, zopiclone or related compounds, including melatonin and melatonin related compounds.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or 5 half-lives prior to the first night of single-blind study medication (whichever was longer).
* Had sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first night of single-blind study medication, or had flown across greater than 3 time zones within 7 days prior to screening.
* Participated in a weight-loss program or had substantially altered their exercise routine within 30 days prior to the first night of single-blind study medication.
* A history of, or currently had, conditions that would affect balance such as:

  * Orthostatic hypotension.
  * Dizziness.
  * Vertigo, or benign paroxysmal positional vertigo.
  * A history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, periodic leg movement syndrome, or fibromyalgia.
* A history of psychiatric disorder (including anxiety, depression, mental retardation, cognitive disorder, bipolar illness and schizophrenia) within the past 6 months.
* A history of drug addiction or drug abuse within the past 12 months.
* A history of alcohol abuse within the past 12 months or regularly consumed more than 14 alcoholic drinks per week or consumed any alcoholic drinks within 24 hours of all polysomnography visits.
* A current significant neurological (including cognitive and psychiatric disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to the first night of single-blind study medication.
* Used tobacco products during nightly awakenings.
* Used melatonin, or other drugs or supplements known to affect sleep/wake function within 1 week or 5 half-lives of the drug (whichever was longer) prior to the first day of single-blind study medication.
* Used any central nervous system (CNS) medication within 1 week or 5 half lives of the drug (whichever was longer) prior to the first day of single-blind study medication.
* Intended to continue taking any disallowed medication or any prescription medication, over the counter (OTC) or herbal medication known to affect the sleep/wake function or otherwise interfere with evaluation of the study medication.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram (ECG), or clinical laboratory tests.
* A positive urine drug screen including alcohol at screening or a positive breathalyzer test at each check-in.
* An apnea hypopnea index (per hour of sleep) >10 as seen on PSG, on the first night of the PSG screening.
* Periodic leg movement with arousal index (per hour of sleep) >10 as seen on PSG, on the first night of PSG screening.
* Any additional condition(s) that in the investigator's opinion would (a) affect sleep/wake function, (b) prohibit the subject from completing the study, or (c) not be in the best interest of the subject.
* Had lower limb prosthetics.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Calculated Area of Center of Pressure (COP) in cm2 recorded on the AccuSway® balance platform during Night 14 with Eyes Open | 1.5 to 2 hours Postdose on Night 14.

SECONDARY OUTCOMES:
Calculated Area of Center of Pressure (COP) in cm2 recorded on the AccuSway® balance platform during Night 14 with Eyes Closed. | 1.5 to 2 hours Postdose on Night 14.
Latency to Persistent Sleep Over a 2-night Average Measured by Polysomnography (Nights 1-2). | Nights 1 and 2.
Latency to Persistent Sleep Over a 2-night Average Measured by Polysomnography (Nights 27-28). | Nights 27 and 28.
Subjective Sleep Latency Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Subjective sleep latency Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Subjective Total Sleep Time Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Subjective Total Sleep Time Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Subjective Wake Time After Sleep Onset Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Subjective Wake Time After Sleep Onset Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Subjective Number of Awakenings Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Subjective Number of Awakenings Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Subjective Sleep Quality Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Subjective Sleep Quality Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Restorative Nature of Sleep Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2.
Restorative nature of sleep Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28.
Morning Alertness Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2
Morning Alertness Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28
Morning Ability to Concentrate Measured by a Post-sleep Questionnaire (Nights 1-2). | Nights 1 and 2
Morning Ability to Concentrate Measured by a Post-sleep Questionnaire (Nights 27-28). | Nights 27 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Principal Investigator — Takeda Global Research & Development Centre (Europe)
Locations (1):
- London, United Kingdom

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI